CLINICAL TRIAL: NCT04763707
Title: Diagnostic Accuracy of Serum Visfatin and Serum Vaspin in Patients With Hepatocellular Carcinoma on Top of Liver Cirrhosis
Brief Title: Serum Visfatin and Serum Vaspin in Patients With Hepatocellular Carcinoma on Top of Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Walaa Abdel Hamed Ali, Diagnostic Accuracy of Serum Visfatin and Serum Vaspin in Patients with Hepatocellular Carcinoma on Top of Liver Cirrhosis, Sohag University
Other Study IDs: Soh-Med-21-02-04
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — serum sample of each participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 : Hepatocellular carcinoma HCC patients with HCV: 40 HCV-related liver cirrhosis patients with HCC on top (Group 1).
- Group 2 : Cirrhotic patients with HCV: 30 HCV-related liver cirrhosis patients(Group 2).
- Group 3 : Healthy control: 20 healthy volunteers will be included as controls(Group 3).

SUMMARY:
Hepatocellular carcinoma (HCC) has a global importance due to its high rate of progression and high mortality rates. Significant risk factors for the development of HCC are metabolic syndrome, obesity and type 2 diabetes mellitus(T2DM). Dysregulation of adipose tissue derived hormones(adipocytokines/adipokines) might also be involved in obesity-related liver carcinogenesis & due to the wide spectrum of visfatin and vaspin activities ,we focus in this study on their potential role in patients with HCV-related liver cirrhosis with and without HCC on top.

DETAILED DESCRIPTION:
Despite improvements in HCC therapy, the prognosis for HCC patients remains poor due to a high incidence of recurrence. Early diagnosis can significantly improve the overall survival of HCC patients. However, currently available diagnostic markers are still inadequate and limited by their low sensitivity and specificity. For instance, the gold standard marker alpha-fetoprotein (AFP) has a false negative rate up to 40% for early stage of HCC. It is worthy to mention that the level of AFP was reported in a normal range of 25% of patients with advanced HCC.

As such, AFP has been excluded from being a marker for the diagnosis of HCC by Practice Guidelines of the American Association for the study of Liver Diseases (AASLD) and confirmed by other studies.

These discrepancies suggest the need of discovering new reliable diagnostic markers for patients with HCC. An improved understanding of the pathogenesis of HCC development would facilitate the development of more effective outcomes for the diagnosis and treatment of HCC at earlier stages.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of CHC will be based on positive HCV antibodies by enzyme-linked immunosorbent assay(ELIZA)& HCV RNA by Polymerase chain reaction ( PCR) for more than 6 months. The diagnosis of liver cirrhosis will be based on clinical data and findings on abdominal ultrasound. The diagnosis of HCC will be based on the typical features of dynamic imaging by triphasic CT with or without elevated serum alpha-fetoprotein (AFP) .

Exclusion Criteria:

* - Co-infection with HBV.
* Presence of clinically suspected other causes of hepatocellular injury ( any history of alcoholism, autoimmune hepatitis, primary sclerosing cholangitis (PSC), primary biliary cholangitis (PBC), Wilson's disease, fatty liver disases with metabolic syndrome &drug induced liver disease.
* Patients diagnosed with other malignancies.
* Patients with history of prior local or systemic HCC-specific treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 70 patients with HCV-related liver cirrhosis attending the outpatient clinic or inpatient section of the department will be included in the study, patients will be categorized into 2 groups:
  * 40 HCV-related liver cirrhosis patients with HCC on top (Group 1).
  * 30 HCV-related liver cirrhosis patients(Group 2).
  * In addition, 20 healthy volunteers will be included as controls(Group 3).
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
serum Visfatin & serum Vaspin levels | they are measured once in all groups then compared after collection of samples, this will be in average 1.5 years
  The 2 markers will be measured in the 3 groups , compared with each one & asses if they are valuable as diagnostic markers for HCC , staging HCC , chronic liver diseases & Metabolic disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Khairy Hammam Morsy, Professor, Study Director — Sohag University
Locations (1):
- Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
we still not decide , due to risk of re-use of data for purposes not approved by participants